CLINICAL TRIAL: NCT05703763
Title: The Applanation Tonometry in Giant Cell Arteritis Pilot
Brief Title: The Applanation Tonometry in GCA Pilot
Acronym: ATOM-GCA
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Jean-Paul Makhzoum, Director - Vasculitis Research Program, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 2020-1890
Record Dates: First submitted 2023-01-17; First posted 2023-01-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Giant Cell Arteritis
Keywords: diagnosis
MeSH Terms: conditions — Giant Cell Arteritis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GCA group: Definite confirmation of GCA will occur 6 months after study inclusion, following the phone follow-up, and will require all the following features: 1) initial symptoms and clinical evolution consistent with GCA; 2) at least one positive test for cranial GCA (ultrasound of temporal arteries, temporal artery biopsy, cranial MRI, cranial PET); and 3) satisfies the 2022 ACR-EULAR classification criteria for GCA.
  Interventions: Diagnostic Test: Applanation tonometry; Diagnostic Test: Standardized GCA assessment; Diagnostic Test: Repeat applanation tonometry (optional)
- Non-GCA group: Participants who do not meet the criteria (above) for GCA at month 6.
  Interventions: Diagnostic Test: Applanation tonometry; Diagnostic Test: Standardized GCA assessment

INTERVENTIONS:
Diagnostic Test: Applanation tonometry — Applanation tonometry will be used to measure arterial stiffness in these segments, bilaterally:
  * Superficial temporal artery to frontal temporal artery
  * Common carotid artery to superficial temporal artery
Diagnostic Test: Standardized GCA assessment — Clinical assessment, blood test review, high-resolution temporal artery ultrasound using a 24mHz probe.
Diagnostic Test: Repeat applanation tonometry (optional) — Repeat index test at month 6 and at disease relapse.
  Groups: GCA group

SUMMARY:
The Applanation Tonometry in Giant Cell Arteritis (ATOM-GCA) study will answer the following questions:

1. How does PWV, measured by applanation tonometry of temporal arteries, differ between patients with and without a final diagnosis of GCA (based on pre-defined criteria 6 months after inclusion)?
2. What is the diagnostic accuracy and positivity cutoff of the PWV, measured by applanation tonometry, in detecting:

   1. A clinical diagnosis of GCA (based on pre-defined criteria 6 months after inclusion)?
   2. Inflammation of temporal arteries on high-resolution ultrasound?
3. What is the acceptability and adherence of repeat applanation tonometry during the follow-up period in patients with GCA?

DETAILED DESCRIPTION:
ATOM-GCA is a single-center, cross-sectional vanguard study.

ELIGIBILITY:
Inclusion criteria:

To be included in ATOM-GCA, participants must meet all the following criteria:

1. Age > 50 years.
2. Referral for suspected, new-onset GCA.
3. Ability to understand and willingness to sign an informed consent form.
4. Willingness to comply with study visits and procedures.

Exclusion criteria:

An individual who meets any of these criteria will be excluded from ATOM-GCA:

1. Referral for a suspected GCA relapse.
2. Current use of systemic glucocorticoids, with the following duration at the baseline visit:

   1. ≥ 14 consecutive days of oral glucocorticoids in the previous 30 days, or
   2. ≥ 7 consecutive days of oral glucocorticoids if intravenous glucocorticoids were administered in the previous 30 days.
3. Current use of any conventional or biologic immunosuppressive therapy.
4. Temporal artery biopsy prior to the study visit.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for suspected new-onset GCA
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
PWV in patients with and without GCA | Baseline
  The primary outcome of ATOM-GCA is to compare the mean PWV in patients with GCA to the mean PWV in individuals without GCA. Final confirmation of GCA will be determined 6 months after study inclusion. This analysis will establish whether the PWV differs in GCA. Additionally, we will explore the optimal PWV cutoff and evaluate its diagnostic performance to confirm a final diagnosis of GCA at 6 months.

SECONDARY OUTCOMES:
Diagnostic performance of the PWV | Baseline
  The secondary outcome is to assess the diagnostic performance of the PWV to predict the presence of GCA-induced inflammation on high-resolution ultrasound. This analysis will identify the optimal PWV cutoff to potentially replace temporal artery ultrasound in GCA diagnosis.

OTHER OUTCOMES:
Proportion of participants who accept repeat applanation tonometry | Baseline
  In patients with GCA, we will evaluate the acceptability of applanation tonometry by measuring the proportion of participants who, at the baseline visit, consent to undergo repeated applanation tonometry during the follow-up period.
Proportion of participants who complete repeated applanation tonometry | Up to 2 years
  The adherence of repeat applanation tonometry (proportion of patient who successfully complete applanation tonometry at month 6 and at relapse) will be assessed in those who consented to have repeat applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Makhzoum, Study Chair — CISSS du Nord-de-l'ile de Montreal
Locations (1):
- Vasculitis Clinic, Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zarka F, Rheaume M, Belhocine M, Goulet M, Febrer G, Mansour AM, Troyanov Y, Starnino T, Meunier RS, Chagnon I, Routhier N, Benard V, Ducharme-Benard S, Ross C, Makhzoum JP. Colour Doppler ultrasound and the giant cell arteritis probability score for the diagnosis of giant cell arteritis: a Canadian single-centre experience. Rheumatol Adv Pract. 2021 Nov 10;5(3):rkab083. doi: 10.1093/rap/rkab083. eCollection 2021. PMID 34859177
- [Background] Baalbaki H, Jalaledin D, Lachance C, Febrer G, Rheaume M, Makhzoum JP. Characterization of visual manifestations and identification of risk factors for permanent vision loss in patients with giant cell arteritis. Clin Rheumatol. 2021 Aug;40(8):3207-3217. doi: 10.1007/s10067-021-05643-5. Epub 2021 Feb 12. PMID 33580374
- See also: Vasculitis Clinic - University of Montreal — http://vasculitemontreal.com